CLINICAL TRIAL: NCT05989347
Title: A Pilot Study to Evaluate Biomarkers and Safety of Dapagliflozin Concomitant with Neoadjuvant Therapy for Patient with HER2-negative Early-stage Breast Cancer and Hyperinsulinemia
Brief Title: Study to Evaluate Biomarkers and Safety of Dapagliflozin Concomitant with Neoadjuvant Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000033529; No NIH funding (Other: 10.18.23)
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Hyperinsulinism; HER2-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Hyperinsulinism | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Women with BMI ≥ 25 kg/m2 and hyperinsulinemia (HOMA-IR ≥ 2.5) and early stage, operable HER2-negative (by FISH or IHC 0, 1+ or 2+) breast cancer for whom systemic neoadjuvant chemotherapy is indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dapagliflozin (Experimental): All participants (with insulin resistance and Estrogen Receptor (ER)+HER2-negative or ER/Progesterone receptor (PR)/HER2-negative breast cancer) will receive current standard of care neoadjuvant chemotherapy as determined by the treating physician, plus dapagliflozin 10 mg orally taken daily throughout chemotherapy treatment.
  Interventions: Drug: Dapagliflozin 10mg

INTERVENTIONS:
Drug: Dapagliflozin 10mg — 10 mg tablets for oral administration daily throughout chemotherapy treatment

SUMMARY:
The primary objective of the study is to assess metabolic plasma markers of insulin resistance in patients with early-stage HER2-negative breast cancers receiving dapagliflozin concomitant with neoadjuvant therapy.

DETAILED DESCRIPTION:
This is a single arm, open label trial that will evaluate changes in plasma markers of insulin resistance, namely, fasting glucose and insulin, measured as the HOMA-IR score, as well as the safety of the addition of dapagliflozin to neoadjuvant treatment in hyperinsulinemic women with newly diagnosed early stage HER2-negative breast cancers who are candidates for neoadjuvant therapy.

Hypotheses are: (i) the SGLT2 inhibitor, dapagliflozin, administered concomitantly with weekly neoadjuvant therapy in hyperinsulinemic women with newly diagnosed HER2-negative breast cancers will lead to a decrease in fasting plasma insulin and glucose and thus, a downregulation in downstream insulin signaling in the tumor as measured by Protein kinase B (PKB)/AKT phosphorylation. (ii) that dapagliflozin can be safely coadministered at full dose with multiagent chemotherapy or chemo-immunotherapy.

Routine, standard of care neoadjuvant chemotherapy, with or without immunotherapy, will be given together with the investigational product. Acceptable chemotherapy regimens include: 1) weekly paclitaxel x12 treatments followed by every two-week doxorubicin, cyclophosphamide (ddAC) x 4 treatments (ddAC-T; ); 2) pembrolizumab every 3 weeks (Q3W), with carboplatin + weekly paclitaxel (cycles 1-4) x12 weeks followed by ddAC x 4 treatments (cycles 5-8) (KEYNOTE-522 regimen; only for participants with stage II-III ER/PR and HER-negative breast cancer); 3) docetaxel plus cyclophosphamide and 4) docetaxel plus carboplatin.

The primary objective of the study is to assess metabolic plasma markers of insulin resistance in participants with early-stage HER2-negative breast cancers receiving dapagliflozin concomitant with neoadjuvant therapy.

Secondary objectives are to assess tissue expression of insulin signaling intermediates and SGLT2 by immunohistochemistry (IHC) on pre- and post-treatment tissue samples.

Outcomes will be assessed before treatment and 12 weeks post treatment (after completion of all neoadjuvant therapy but before surgery).

Registration (including outcome measures) was updated to reflect current protocol July 2024.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years of age with newly diagnosed, histologically confirmed, clinical stage I-III, HER2-negative - either ER+ or triple negative - invasive breast cancer as defined by ASCO CAP guidelines for whom neoadjuvant chemotherapy would be indicated. The following chemotherapy regimens are acceptable:

  1. Weekly or dose dense paclitaxel, followed by dose dense doxorubicin plus cyclophosphamide
  2. Docetaxel plus cyclophosphamide
  3. Docetaxel plus carboplatin plus or minus pembrolizumab
  4. Paclitaxel plus carboplatin concurrent with every 3 week pembrolizumab followed by dose dense doxorubicin plus cyclophosphamide concurrent with every 3 week pembrolizumab (KEYNOTE-522 regimen; only for participants with triple negative breast cancer)
* BMI ≥ 25 kg/m2
* Hyperinsulinemia defined as HOMA-IR ≥ 2.5.
* Willing and able to provide written informed consent for the trial.
* Has at least one (1) physical 4-5-micron single H&E slide from diagnostic biopsy available
* Female participants of childbearing potential should have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female participants must be 1 year post-menopausal orsurgically sterile, Women of childbearing potential who are sexually active with a non-sterilized male partner must agree to follow their chemotherapy provider's instructions for birth control.
* Participants should have adequate organ function to tolerate chemotherapy, as defined by:

  1. peripheral granulocyte count of > 1,500/mm3
  2. platelet count > 100,000/mm3
  3. hemoglobin >9 g/dL
  4. total bilirubin < 1.5 x upper limit of normal (ULN)
  5. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) each < 1.5 x ULN
  6. serum creatinine < 1.5 x ULN
  7. INR/PT/PTT each < 1.5 x ULN
* Able to swallow oral formulation of the study agent
* Subjects should not donate blood while participating in this study, or for at least 90 days following the last dose of chemotherapy

Exclusion Criteria:

* Participants who underwent partial excisional biopsy or lumpectomy, segmental mastectomy or modified radical mastectomy or sentinel node biopsy and therefore cannot be assessed accurately for pathologic response, are not eligible.
* Participants currently pregnant or breastfeeding.
* Participants for whom any of the planned chemotherapies are contraindicated.
* Participants with currently diagnosed type I or II diabetes mellitus.
* Participants taking any antidiabetic medication that would affect insulin resistance or hyperinsulinemia (i.e. TZD, GLP-1RA, DPP-4i, SGLT2i, metformin) in the past one month.
* Participants with history of hypersensitivity reaction to dapagliflozin.
* Participants with eGFR < 25.
* History of recurrent (three or more occurrences within 12 months, or two or more occurrences within 6 months) urinary tract infections.
* Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight) or have a history of gastrointestinal surgery.
* Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, intranasal influenza, rabies, BCG, and typhoid vaccine.
* Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) | baseline, post paclitaxel treatment at week 12, and 2 weeks post neoadjuvant therapy
  Change in HOMA-IR (calculated as fasting insulin (μU/ml) x fasting glucose (mmol/l) divided by 22.5.

SECONDARY OUTCOMES:
Change in Fasting glucose concentration | baseline, post paclitaxel treatment at week 12, and 2 weeks post neoadjuvant therapy
  Fasting plasma glucose concentration will be assessed following an overnight fast at baseline and 12 weeks post treatment
Change in Fasting insulin concentration | baseline, post paclitaxel treatment at week 12, and 2 weeks post neoadjuvant therapy
  Fasting plasma insulin concentration will be assessed at baseline and 12 weeks post treatment
Total and phosphorylated PKB/AKT | baseline, post paclitaxel treatment at week 12, and 2 weeks post neoadjuvant therapy
  Immunohistochemistry (IHC) staining for expression of Total and phosphorylated PKB/AKT in breast cancer tissue, before and after (in participants with residual cancer) treatment. For quantification of IHC, sections will be scored manually by a pathologist using the Allred system, a clinical instrument based on the percentage of cells that stain by immunohistochemistry for PKB/AKT (on a scale of 0 to 5) and the intensity of that staining (on a scale of 0 to 3, for a possible maximum total score of 8. The lower the number the less staining.
Total and phosphorylated insulin receptor | baseline, post paclitaxel treatment at week 12, and 2 weeks post neoadjuvant therapy
  Immunohistochemistry (IHC) staining for expression of Total and phosphorylated insulin receptor in breast cancer tissue, before and after (in participants with residual cancer) treatment. For quantification of IHC, sections will be scored manually by a pathologist using the Allred system, a clinical instrument based on the percentage of cells that stain by immunohistochemistry for PKB/AKT (on a scale of 0 to 5) and the intensity of that staining (on a scale of 0 to 3, for a possible maximum total score of 8. The lower the number the less staining.
Total and phosphorylated insulin-like growth factor-1 receptor (IGF1R) | baseline, post paclitaxel treatment at week 12, and 2 weeks post neoadjuvant therapy
  Immunohistochemistry (IHC) staining for expression of Total and phosphorylated insulin-like growth factor-1 receptor (IGF1R) in breast cancer tissue, before and after (in participants with residual cancer) treatment. For quantification of IHC, sections will be scored manually by a pathologist using the Allred system, a clinical instrument based on the percentage of cells that stain by immunohistochemistry for PKB/AKT (on a scale of 0 to 5) and the intensity of that staining (on a scale of 0 to 3, for a possible maximum total score of 8. The lower the number the less staining.
Total and phosphorylated insulin receptor substrate (IRS) 1 | baseline, post paclitaxel treatment at week 12, and 2 weeks post neoadjuvant therapy
  Immunohistochemistry (IHC) staining for expression of Total and phosphorylated insulin receptor substrate (IRS) 1 in breast cancer tissue, before and after (in participants with residual cancer) treatment. For quantification of IHC, sections will be scored manually by a pathologist using the Allred system, a clinical instrument based on the percentage of cells that stain by immunohistochemistry for PKB/AKT (on a scale of 0 to 5) and the intensity of that staining (on a scale of 0 to 3, for a possible maximum total score of 8. The lower the number the less staining.
Sodium-glucose cotransporter-2 (SGLT2) | baseline, post paclitaxel treatment at week 12, and 2 weeks post neoadjuvant therapy
  Immunohistochemistry (IHC) staining for expression of SGLT2 in breast cancer tissue, before and after (in participants with residual cancer) treatment. For quantification of IHC, sections will be scored manually by a pathologist using the Allred system, a clinical instrument based on the percentage of cells that stain by immunohistochemistry for PKB/AKT (on a scale of 0 to 5) and the intensity of that staining (on a scale of 0 to 3, for a possible maximum total score of 8. The lower the number the less staining.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Lustberg, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center Smilow Cancer Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No